CLINICAL TRIAL: NCT00000769
Title: A Phase I/II Study of Recombinant Interleukin-4 in AIDS and Kaposi's Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 224; 11201 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome; Interleukin-4
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Interleukin-4

INTERVENTIONS:
Drug: Interleukin-4

SUMMARY:
To determine the safety and tolerance of interleukin-4 (IL-4) in patients with AIDS-related Kaposi's sarcoma. To determine the effects of IL-4 on tumor growth in patients with AIDS-related Kaposi's sarcoma.

IL-4 exhibits a variety of beneficial effects on the immune system and is a potent inhibitor of Kaposi's sarcoma cells in vitro.

DETAILED DESCRIPTION:
IL-4 exhibits a variety of beneficial effects on the immune system and is a potent inhibitor of Kaposi's sarcoma cells in vitro.

Patients are stratified into two groups according to CD4 count (less than 100 cells/mm3 and greater than or equal to 100 cells/mm3) and are enrolled in cohorts of four patients at each of four dose levels of IL-4 per stratum. Within each stratum, if patients at a given dose level have received at least 2 weeks of study therapy and no more than two patients experienced grade 3 or 4 drug-related toxicity, dose escalation in subsequent patients may begin. The MTD is defined as the dose at which 50 percent of patients develop grade 3 or worse toxicity. Patients with CD4 count less than 500 cells/mm3 (per 12/30/94 amendment) must be on antiretroviral therapy during study treatment.

PER AMENDMENT 11/20/95: Group I - enrollment is closed, the objective has been defined. Group II - patients must have CD4 cells greater than or equal to 100/mm3 and less than 500/mm3.

PER AMENDMENT 11/20/95: All patients will receive antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Antiretroviral therapy during study treatment only in patients with CD4 count < 500 cells/mm3 (per 12/30/94 amendment).

Allowed:

* G-CSF for a second occurrence of grade 3 or 4 neutropenia (per 12/30/94 amendment).
* Nonsteroidal anti-inflammatory agents including acetaminophen for drug-related fevers.
* Systemic steroids for no more than 1 week in any 30-day period.
* PCP prophylaxis with TMP/SMX, dapsone, or inhaled pentamidine, if patient has a history of PCP or a CD4 count < 250 cells/mm3.

Allowed only in patients with CD4 count < 100 cells/mm3:

* Maintenance doses of ganciclovir, pyrimethamine/sulfa and TMP/SMX for stable, well-controlled opportunistic infections.
* Non-myelosuppressive treatment IND medications.

Prior Medication: Required: PER AMENDMENT 11/20/95:

* Stable dose of antiretroviral therapy required for at least 21 days prior to study entry for all patients. (Changed from - Stable dose of antiretroviral therapy for at least 21 days prior to study entry in patients with CD4 count < 500 cells/mm3 (per 12/30/94 amendment).

Patients must have:

* AIDS-related Kaposi's sarcoma.
* PER AMENDMENT 11/20/95: CD4 lymphocyte count >= 100 but < 500 cells/mm3. (Changed from - HIV infection.)
* PER AMENDMENT 11/20/95: All Patients will receive antiretroviral therapy. (Changed from - Current antiretroviral therapy IF CD4 count < 500 cells/mm3 (per 12/30/94 amendment).)
* No active opportunistic infections requiring induction therapy.
* Consent of parent or guardian if less than 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Other active malignancies (except basal cell carcinoma of the skin and in situ cervical cancer).
* Alteration in mental status that may prevent compliance.
* Cardiac functional capacity of Class II or worse OR regional wall abnormalities or abnormal ejection fraction on two-dimensional echocardiogram, if performed.

Concurrent Medication:

Excluded:

* Chemotherapy, interferons, or immune modulators for Kaposi's sarcoma.
* Myelosuppressive agents such as induction doses of ganciclovir, Fansidar (pyrimethamine/sulfadoxine), or any other investigational drugs (with the exception of non-myelosuppressive treatment IND medications in specific patients).
* GM-CSF or erythropoietin (except for a second grade 3/4 neutropenia or anemia).
* G-CSF.

Patients with the following prior conditions are excluded:

* History of myocardial infarction or significant arrhythmias.
* History of symptomatic hypoglycemia.

Prior Medication:

Excluded:

* Systemic therapy (including chemotherapy, interferons, and immune modulators) for Kaposi's sarcoma within 4 weeks prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48
Dates: Study Completion 1998-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miles S, Study Chair; Scadden D, Study Chair
Locations (3):
- United States (3):
  - UCLA CARE Center CRS, Los Angeles, California
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts

REFERENCES:
- [Background] Miles SA, Mitsuyasu R, LaFleur F, Ryback M, Kasden P, Suckow C, Groopman J, Scadden D. Phase I/II trial of interleukin-4 in KS (ACTG 224). Int Conf AIDS. 1994 Aug 7-12;10(1):46 (abstract no 159B)